

C.I. EOM-28-21

#### CEIm Fundació Sant Joan de Déu

# DICTAMEN DEL COMITÉ DE ÉTICA DE LA INVESTIGACIÓN CON MEDICAMENTOS

Dr. Jesús Pineda Sánchez Presidente del CEIm Fundació Sant Joan de Déu

#### **HACE CONSTAR:**

Que el CEIm Fundació Sant Joan de Déu en su reunión del día **15/09/2022**, acta **16/2022**, ha evaluado la propuesta del promotor sobre la **Modificación sustancial nº 1** referida al estudio:

**Título:** "Estudio de hipersensibilidad a Anti-Inflamatorios No Esteroideos (AINES) en población

pediátrica"

Investigador Principal: Adrianna Machinena Spera

Código CEIm: EOM-28-21

Servicio: Alergia e immunología clínica

Centro: Hospital Sant Joan de Déu - Esplugues HSJD.1 (FSJD)

### **Documentos con versiones:**

| Protocolo | Versión 2, agosto 2022 |
|---|---|
| Hoja de información al paciente /padre o tutor legal | Versión 2, agosto 2022 |
| Hoja de consentimiento de los padres o tutor legal del<br>menor participante (utilizar en estudios en los que<br>participe un menor de 18 años) | Versión 2, agosto 2022 |
| Hoja de información y asentimiento al paciente | Versión 2, agosto 2022 |

Que este CEIm considera que no se aumenta el riesgo de los pacientes y que se pueden cumplir las finalidades del estudio por lo que emite un **INFORME FAVORABLE** para la realización de la modificación anteriormente mencionada.

Que el CEIm Fundació Sant Joan de Déu, tanto en su composición, como en los PNT cumple con las normas de BPC (CPMP/ICH/135/95); se cumplieron los requisitos establecidos en la legislación vigente - Real Decreto 1090/2015 - para que la decisión del citado CEIm sea válida; su composición actual es la siguiente:

| Presidente | Dr. Jesús Pineda Sánchez (Medicina - Pediatría) |
|--------------------|---------------------------------------------------|
| Vicepresidente | Dr. Bernabé Robles (Medicina – Neurología) |
| Secretaria técnica | Dra. Neus Riba Garcia (Farmacología Clínica) |
| Vocales | Hno. Fernando Aguiló Martinez (Medicina Tropical) |
| | Sra. Clara Chamorro Pérez (Jurista) |

C.I. EOM-28-21 Página 1 de 2



C.I. EOM-28-21

## CEIm Fundació Sant Joan de Déu

| Sr. Ángel del Campo Escota (Representante de las asociaciones de pacientes) |
|-----------------------------------------------------------------------------|
| Dra. Beatriz del Pino Gaya (Farmacia hospitalaria) |
| Dr. Pau Ferrer Salvans (Farmacología Clínica) |
| Dra. Ana Maria Martin Ancel (Medicina – Neonatología) |
| Dra. Laura Martínez Rodríguez (Enfermería) |
| Sr. Eduard Puig Vaquero (Jurista – Delegado protección de datos) |
| Sra. María Eugenia Rey Abella (Farmacia AP) |
| Dra. Marisa Serra Alacid (Medicina – Unidad Atención al Usuario) |
| Dra. Rosa María Dueñas (Medicina-Psiquiatra) |
| Dra. Carlota Romans Ruíz (Farmacòleg Clínic-Metge psiquiatra) |
| Dr. Antoni Noguera Julián (Medicina – Pediatria) |
| Dra. Edurne Mazarico Gallego (Medicina – Ginecologia i Obstetrícia) |
| Dra. Esther Via Virgili (Medicina – Psiquiatria) |
| Dr. Oriol Martín Solé (Cirugía y miembro del CR) |
| Dra. Maite Begoña Gorostegui Obanos – (Medicina – Oncología) |

<sup>\*\*</sup>En el caso de que se evalúe algún proyecto del que un miembro sea investigador/colaborador, este se ausenta de la reunión durante la discusión del proyecto.

Para que conste donde proceda, y a petición del promotor,

Lo que firmo en Esplugues de Llobregat (Barcelona), a

Fdo:

Dr. Jesús Pineda Sánchez Presidente del CEIm Fundació Sant Joan de Déu

C.I. EOM-28-21 Página 2 de 2